CLINICAL TRIAL: NCT06924762
Title: Efficacy and Safety of Interleukin-2 Treatment in Moderate to Severe Chronic Spontaneous Urticaria With Poor Control by Antihistamines: a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Interleukin-2 for Refractory Chronic Spontaneous Urticaria
Acronym: ESIT-CSU
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Tongji Hospital (Other); West China Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Fujian Medical University Union Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The First People's Hospital of Changde City (Other); The Third People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Hai Long, M.D., Ph.D. & Vice President, The Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYG20240044; MR-43-25-003708 (Other: Chinese Clinical Trial Registry (ChiCTR))
Record Dates: First submitted 2024-11-24; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Chronic Spontaneous Uriticaria
Keywords: Interleukin-2; Chronic spontaneous uriticaria; urticaria control test; poor response to second-generation antihistamines
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled, parallel group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interleukin-2 treatment group (Experimental): The enrolled subjects will receive three cycles of interleukin-2 treatment in the first 12 weeks upon initiation of the intervention, while continuing with the same oral regimen of second-generation antihistamines as they have been receiving before initiation of the trial. In each cycle of interleukin-2 treatment, the enrolled subjects will receive an intramuscular injection of interleukin-2 at a dosage of 1 million international units, dissolved in 1.0 mL of sterile water for injection, once daily for 7 consecutive days. The three cycles of interleukin-2 treatment will be administered on Day 0~6, Day 28~34 and Day 56~62, respectively.
  Interventions: Drug: Human interleukin-2 (I) intramuscular injection
- Placebo group (Placebo Comparator): The enrolled subjects will receive three cycles of placebo injections in the first 12 weeks upon initiation of the intervention, while continuing with the same oral regimen of second-generation antihistamines as they have been receiving before initiation of the trial. In each cycle of placebo injections, the enrolled subjects will receive an intramuscular injection of placebo at a same specification as in the IL-2 treatment group, dissolved in 1.0 mL of sterile water for injection, once daily for 7 consecutive days. The three cycles of placebo injections will be administered on Day 0~6, Day 28~34 and Day 56~62, respectively.
  Interventions: Drug: Placebo intramuscular injection

INTERVENTIONS:
Drug: Placebo intramuscular injection — On the basis of background treatment, intramuscular injection of placebo was added.
  Arms: Placebo group
Drug: Human interleukin-2 (I) intramuscular injection — On the basis of background treatment, intramuscular injection of human interleukin-2 (I) will be added.
  Arms: Interleukin-2 treatment group

SUMMARY:
The goal of this clinical trial is to learn if human interleukin-2 (IL-2) works to treat moderate to severe chronic spontaneous urticaria in adults who remain symptomatic despite oral antihistamine treatment (refractory CSU). It will also learn about the safety of IL-2. The main questions it aims to answer are:

Does IL-2 alleviate the symptoms of urticaria in patients? What medical problems do participants have when given IL-2? Researchers will compare IL-2 to a placebo (a look-alike and smell-like substance that contains no IL-2) to see if IL-2 works to treat refractory, moderate to severe CSU.

Participants will:

Receive IL-2 or a placebo intramuscular injections for 3 rounds at Week 0, 4 and 8, in which each round includes one injection daily for seven consecutive days.

Visit the clinic for checkups and tests at Week 2, 4, 8, 12 and 24. Keep a diary of their symptoms and the number of tablets of oral antihistamines.

DETAILED DESCRIPTION:
Background:

Urticaria is a common disorder characterized by localized edema due to dilation and increased permeability of small blood vessels in the skin and mucous membranes. The primary clinical manifestations include wheals and pruritus.

Chronic spontaneous urticaria (CSU) is defined as recurrent, transient (<24 hours), pruritic wheals on the skin and mucosa lasting for more than 6 weeks, with or without angioedema, excluding chronic inducible urticaria. Among patients with chronic urticaria, about 2/3 have CSU. Although the pathogenesis of CSU remains unclear, increasing evidence suggests an autoimmune feature of this disorder. Oral antihistamines are the primary treatment for CSU, yet some patients continue to experience symptoms despite treatment with standard or double doses. Recent studies have shown that human IL-2 (Interleukin-2) can be effective in a proportion of CSU patients refractory to antihistamine treatment, without significant side effects. Therefore, in this clinical trial we aim to evaluate the therapeutic effect and safety of this new therapeutic method.

Study Design:

This is a randomized, placebo-controlled, multi-center clinical trial to evaluate the safety and efficacy of IL-2 treatment in CSU patients who remain symptomatic despite oral antihistamine treatment.

Methods:

CSU patients who meet the inclusion criteria will receive IL-2 or placebo intramuscular injections in combination with their current antihistamine regimen (either a single antihistamine or a combination of two to three antihistamines at a dose of at least the standard dosage). Endpoints include clinical response, quality of life, and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Not limited; Age: at least 18 years old and less than 75 years old;
2. Diagnosed with chronic spontaneous urticaria (CSU) (including patients overlapped with chronic inducible urticaria) according to the 2021 EAACI/GA²LEN/EDF/AAAAI guidelines;
3. Disease course of CSU for at least 12 weeks;
4. The patient has been treated with second-generation antihistamines (one or more types, up to 4 tablets per day) every day for 2 weeks or more but still experiences significant symptoms of wheals and/or itching, with a UAS7 score ≥16 or a UCT score <12;
5. UAS7 ≥16 on the date prior to randomization (according to complete daily symptom log data recorded in the past 7 days before randomization);
6. Willing and able to complete daily symptom logs throughout the entire study period;
7. The patient voluntarily consents to participate in this research project and has signed the informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women, or women planning to conceive within 6 months;
* Has used corticosteroids, immunosuppressants, leukotriene receptor antagonists, H2 receptor antagonists, intravenous immunoglobulin (IVIG) therapy, and/or undergone plasma exchange in the past 4 weeks;
* Has received omalizumab or other biologic treatments in the past 12 weeks;
* Has previously undergone interleukin-2 treatment;
* Has a history of anaphylactic shock;
* Plans or anticipates the use of any prohibited drugs or treatments during the screening and/or treatment periods;
* Currently has active or recurrent severe infections, such as active tuberculosis;
* Has a congenital or acquired immunodeficiency disorder;
* Has a history of drug or alcohol abuse, mental disorders, or poor compliance, making them unable to adhere to treatment;
* Currently enrolled in another clinical trial;
* Is an employee of the clinical research facility or directly involved in the study, or is an immediate family member of such an individual;
* Any other reason that makes participation in this trial inappropriate.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Urticaria Activity Score of 7 Days（UAS7）at 12 Weeks | Baseline and 12 weeks.
  This rating requires patients to record the number of wheals and the severity of itching once a day. The sum of each day's UAS score in the past seven consecutive days is UAS7.

SECONDARY OUTCOMES:
Proportion of patients who achieve the treatment target at 2, 4, 8, 12 and 24 weeks, respectively | 2, 4, 8, 12 and 24 weeks post-intervention
  According to the Expert Consensus on Treat⁃To⁃Target in Chronic Spontaneous Urticaria (2023), published in Chinese Journal of Dermatology, we count the proportion of CSU patients who achieve treatment targets at 2, 4, 8, 12 and 24 weeks post IL-2 or placebo intervention. As stated in Table 1 in the Expert Consensus mentioned above, a CSU patient achieves the treatment target when he meets the following criteria: (1) at 2 weeks post-intervention: UAS7 ≤6, or UAS7 decreased by ≥11 from baseline, or chronic urticaria quality of life questionnaire (CU-Q2oL) score increased by ≥8 from baseline; (2) at 4 weeks or 8 weeks: urticaria control test (UCT) score ≥12, or UAS7 ≤6, or UAS7 decreased by ≥11 from baseline, or CU-Q2oL increased by ≥8 from baseline; (3) at 12 weeks: UCT ≥12, or UAS7 ≤6, or CU-Q2oL increased by ≥19 from baseline; (4) at 24 weeks: UCT =16, or UAS7 =0, or CU-Q2oL increased by ≥19 from baseline.
The change from baseline in UAS7 at 2 weeks and 24 weeks, respectively | Baseline, 2 weeks, and 24 weeks
  This rating requires patients to record the number of wheals and the severity of itching once a day. The sum of the wheal score (range 0-3 points; 0 points refer to no wheals in the day, 1 point refers to ≤ 20 wheals, 2 points refer to 20-50 wheals, and 3 points refer to ≥ 50 wheals in the day) and itching score (range 0-3 points; 0 points=none, 1 point=mild itching, 2 points=moderate itching, 3 points=severe itching) is the UAS score for the day. The sum of scores for seven consecutive days is UAS7.
Change from baseline in HSS7 score at 2, 12 and 24 weeks, respectively | Baseline, 2 weeks, 12 weeks and 24 weeks
  This rating requires patients to record the number of wheals once daily. The sum of each day's wheal score (range 0-3 points; 0 points refer to no wheals in the day, 1 point refers to ≤ 20 wheals, 2 points refer to 20-50 wheals, and 3 points refer to ≥ 50 wheals in the day) in the past seven consecutive days is HSS7.
Change from baseline in ISS7 score at 2, 12 and 24 weeks, respectively | Baseline, 2, 12 and 24 weeks
  This rating requires patients to record the severity of itching once a day. The sum of the itching scores (range 0-3 points; 0 points=none, 1 point=mild itching, 2 points=moderate itching, 3 points=severe itching) in the past seven consecutive days is ISS7.
Change from baseline in Dermatology Life Quality Index (DLQI) from baseline at 2, 12 and 24 weeks, respectively | Baseline, 2, 12 and 24 weeks
  DLQI has a total of 10 questions, covering symptoms and feelings, daily activities, leisure and entertainment, work and study, interpersonal relationships, and treatment. The score range for each item is 0-3 points. Those who answer no or irrelevant questions will receive 0 points, while those who answer a lot will receive 3 points. The sum of the scores for each question is the total score (ranging from 0 to 30).
Proportion of CSU patients with no disease activity (UAS7=0) and those with low disease activity (UAS7 ≤6) at 2, 12 and 24 weeks, respectively | Baseline, 2, 12 and 24 weeks
  At each time point (2, 12 and 24 weeks post-intervention), the proportion of CSU patients with UAS7 =0 and the proportion of CSU patients with UAS7 ≤6 are counted, respectively.
Proportion of well-controlled CSU patients (UCT ≥12) and completely controlled CSU patients (UCT=16) at 2, 12 and 24 weeks, respectively | Baseline, 2, 12 and 24 weeks
  At each time point (2, 12 and 24 weeks post-intervention), the proportion of CSU patients with UCT ≥12 and the proportion of CSU patients with UCT =16 are counted, respectively.
Total number of second-generation antihistamines taken per week at 2, 12 and 24 weeks, respectively | Baseline, 2, 12 and 24 weeks
  Record the number of second-generation antihistamines tablets/capsules taken by the patient on a daily basis, and add up the number of pills taken each day in the past seven consecutive days to obtain the total number of second-generation antihistamines taken in the previous week.
Proportion of CSU patients receiving systemic corticosteroid treatment and the total duration of systemic corticosteroid treatment during the study | 24 weeks post-intervention or the date of patient withdrawal from the group
  Record the initiation date and cease date of systemic corticosteroid treatment for each subject since their enrollment in interleukin-2/placebo intervention and calculate the duration (dates). The number of subjects who received systemic corticosteroid treatment during the study was calculated, and the total duration (dates) of systemic corticosteroid treatment was summed up in each group.
Incidence of Adverse Events | 12 and 24 weeks
  Any adverse event is recorded for each subject during the study. Incidence of adverse events, either in total or in separate types of adverse events, is calculated for each treatment group.
Incidence of Severe Adverse Events | 2, 12 and 24 weeks post-intervention
  The ratio of the number of cases with severe adverse events to the total number of cases in each treatment group is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Long, MD, PhD, Principal Investigator — Second Xiangya Hospital of Central South University; Qianjin Lu, MD, PhD, Study Director — Second Xiangya Hospital of Central South University
Locations (1):
- the Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
We would agree to share all IPD collected throughout the trial, but we have not made a decision on this, because we are not sure how to share or by which website we can share this information.